CLINICAL TRIAL: NCT03455933
Title: Action Mechanisms Responsibles for the Effects of Shock Waves on the Pressure Pain Thresholds
Brief Title: Action Mechanisms of Shock Waves on Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Ibai López de Uralde Villanueva, Clinical Professor and Principal Investigator, Centro Universitario La Salle
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CSEU La Salle
Record Dates: First submitted 2018-01-19; First posted 2018-03-07 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Asymptomatic Condition
MeSH Terms: conditions — Asymptomatic Diseases | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Shockwave Light Pain Group (Experimental): Sham Comparator. It will received a light intensity shockwave in the lateral epicondyle regulated until reach a 3/10 in the Visual Analog Scale (VAS) scale.
  Interventions: Other: Sham Comparator
- Shockwave Moderate Pain Group (Experimental): Experimental Intervention. It will received a moderate intensity shockwave in the lateral epicondyle regulated until reach a 6/10 in the Visual Analog Scale (VAS) scale.
  Interventions: Other: Experimental Intervention
- Cold Pressure Group (Other): Control Group. The cold pressure test will be apply to this group. The investigators will use a container with an outer part filled with ice and an inner part filled with water, both separated by a screen that prevents direct contact between the ice and the hand. The water will be regularly stirred to maintain the temperature near to 0.7ºC.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Sham Comparator — The investigators will apply a light intensity shockwave in the lateral epicondyle with the portable SHOCKMASTER 300 at a 8Hz frequency and 2000 impulses. The intensity will be regulated to reach a 3/10 in the VAS scale, depending on the tolerance of the subject. Each patient will receive between 5 and 10 impulses starting with the lower intensity of the device (middle energy: 1 bar) and will go up towards the target (3/10 in VAS).
  Arms: Shockwave Light Pain Group
Other: Experimental Intervention — The investigators will apply a moderate intensity shockwave in the lateral epicondyle with the portable SHOCKMASTER 300 at a 8Hz frequency and 2000 impulses. The intensity will be regulated to reach a 6/10 in the VAS scale, depending on the tolerance of the subject. Each patient will receive between 5 and 10 impulses starting with the lower intensity of the device (middle energy: 1 bar) and will go up towards the target (6/10 in VAS).
  Arms: Shockwave Moderate Pain Group
Other: Control Group — Patients will place their hand, wide open and up to the wrist, into the inner part of the container and will keep it under water for a maximum time of 2 minutes. If pain is unbearable before the time ends, the participant will be able to withdraw the hand.
  Arms: Cold Pressure Group

SUMMARY:
The aim of this study is to evaluate whether the intensity of pain perceived during the application of extracorporeal shockwave therapy (ESWT) is determinant for producing changes in pressure pain threshold (PPT) in asymptomatic subjects. The investigators will perform a single controlled random trial to three groups. Two of them will receive ESWT whereas the third group will get a cold pressure test (CPT).

ELIGIBILITY:
Inclusion Criteria:

* Absence of pain or illness
* No changes in cognitive ability
* Good command of Spanish, both spoken and written

Exclusion Criteria:

* People with systemic diseases, tumors, infections, pacemakers, clotting disorders, skeletally immature, fibromyalgia, whiplash history, dizziness or in physiotherapeutic or pharmacological treatment
* Pregnant women

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold | through study completion, an average of 1 month
  The investigators will use a digital algometer (Force Ten FDX Wagner) to measure when pressure becomes pain.

OTHER OUTCOMES:
Pain Catastrophizing | Baseline
  The Spanish version of the Pain Catastrophizing Scale (PCS) assesses the degree of pain catastrophizing. It assess three components of catastrophizing: rumination, magnification, and helplessness. The PCS is composed of 13 items, which must be answered by a numeric value between 0 (not at all) and 4 (all the time), having a maximum score of 52 points (higher scores indicates more catastrophizing). PCS is a reliable and valid measure of pain catastrophizing (D'Eon JL, Harris CA, Ellis JA. Testing factorial validity and gender invariance of the pain catastrophizing scale. J Behav Med 2004; 27:361-372) (Olmedilla Zafra A, Ortega Toro E, Cano LA. Validation of the Pain Catastrophizing Scale in Spanish athletes. Cuad Psicol del Deport 2013; 13:83-93.).
Kinesiophobia level | Baseline
  Pain-related fear of movement was assessed using the 11-item Spanish version of the Tampa Scale of Kinesiophobia (TSK-11), whose reliability and validity have been demonstrated (Gómez-Pérez L, López-Martínez AE, Ruiz-Párraga GT. Psychometric properties of the Spanish version of the Tampa Scale for Kinesiophobia (TSK). J Pain 2011; 12:425-435.). Each item is scored using a 4-point scale (1 = strongly disagree; 4 = strongly agree). The final score can range between 11 and 44 points, with higher scores indicating greater perceived kinesiophobia
Pain intensity | During the intervention
  Pain intensity was measured with the Visual Analog Scale (VAS). It is a single-item and continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. For pain intensity, as in this study, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]). To avoid clustering of scores around a preferred numeric value, numbers or verbal descriptors at intermediate points are not recommended. The VAS is a reliable and valid measure of pain (Jensen MP, Turner JA, Romano JM, Fisher LD. Comparative reliability and validity of chronic pain intensity measures.Pain 1999; 83:157-162.) (Katz J, Melzack R. Measurement of pain.Surg Clin North Am 1999; 79:231-252.)

CONTACTS AND LOCATIONS:
Overall Officials: Ibai Lopez de Uralde Villanueva, Principal Investigator — Universidad La Salle, Mexico
Locations (1):
- CSEU La Salle Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garcia-Muntion A, Godefroy L, Robert H, Munoz-Garcia D, Calvo-Lobo C, Lopez-de-Uralde-Villanueva I. Study of the mechanisms of action of the hypoalgesic effect of pressure under shock waves application: A randomised controlled trial. Complement Ther Med. 2019 Feb;42:332-339. doi: 10.1016/j.ctim.2018.12.012. Epub 2018 Dec 18. PMID 30670263